CLINICAL TRIAL: NCT04540822
Title: Peripheral Catheter Pressure Ulcer Prevention in Pediatry : Use of Compresses Versus Standard Care"
Brief Title: Peripheral Catheter Pressure Ulcer Prevention in Pediatry : Use of Compresses Versus Standard Care
Acronym: KTESCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHD194-19
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Pressure Ulcer
Keywords: pediatrics; pressure ulcer; peripheral venous catheter
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The childcare assistant in charge of primary outcome assessment should not having taken care of the child before. In addition, the catheter-extension tube junction, with or without compress,will be secured by placing a crepe bandage. The nurse will call him to assess the primary outcome after the catheter ( and compress and crepe bandage) will have been removed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peripheral venous catheter with compress (Experimental): Insertion of a peripheral venous catheter with a compress inserted below the catheter-extension tube junction
  Interventions: Other: peripheral venous catheter with compress under the catheter-extension tube junction
- peripheral venous catheter without compress (Active Comparator): Insertion of a peripheral venous catheter without any compress inserted below the catheter-extension tube junction.
  Interventions: Other: peripheral venous catheter without compress under the catheter-extension tube junction

INTERVENTIONS:
Other: peripheral venous catheter with compress under the catheter-extension tube junction — Placement of a BD Insyte® type catheter of 20 to 24 Gauge calibre on a peripheral vein located in the crease of the elbow or top of the hand or scalp or top of the foot. The catheter is placed while respecting the detersion and disinfection of the skin with the appropriate products and according to the procedure in force in the department. Once the venous return has been checked, a 10 cm extension with a BECTON-DIC® 3-way valve will be connected, which is previously purged with 0.9% Sodium Chloride. Under the catheter-extension tube junction will be inserted a sterile non-woven compress, cut sterilely (3.5x1.5 cm). The assembly will be held in place by a transparent sterile semi-permeable adhesive dressing such as Tegaderm® (5x7 cm). This area will be secured by placing a crepe bandage (crepe bandage 4 m x7 cm).
  Arms: peripheral venous catheter with compress
Other: peripheral venous catheter without compress under the catheter-extension tube junction — Placement of a BD Insyte® type catheter of 20 to 24 Gauge calibre on a peripheral vein located in the crease of the elbow or top of the hand or scalp or top of the foot. The catheter is placed while respecting the detersion and disinfection of the skin with the appropriate products and according to the procedure in force in the department. Once the venous return has been checked, a 10 cm extension with a BECTON-DIC® 3-way valve will be connected, which is previously purged with 0.9% Sodium Chloride. No compresses will be inserted under the catheter-extension tube junction.The assembly will be held in place by a transparent sterile semi-permeable adhesive dressing such as Tegaderm® (5x7 cm). This area will be secured by placing a crepe bandage (crepe bandage 4 m x7 cm).
  Arms: peripheral venous catheter without compress

SUMMARY:
Peripheral venous catheterisation is a multi-daily practice in a paediatric ward.

In our pediatrics department, nurses have observed for several years now the appearance of pressure sore-like skin lesions at the junction of the peripheral venous catheter with the extension tube. A ward habit has spontaneously developed of applying a compress under this junction. The objective is to minimize physical or emotional aggression as well as pain. Pain that is denied or not identified and not relieved is memorized by the child, which can have consequences on the perception of pain and the subsequent acceptance of care.

To date, through their reading and research, investigators have been able to find articles mentioning the risks of pressure ulcers in children related to medical devices. However, few elements are developed concerning catheter-related pressure ulcers, especially on this specific technique for preventing injuries at the catheter-extension tube junction. Investigators have not found any recommendations on this subject.

Thus, the aim of this study is to compare two peripheral venous catheter fixation devices, with compress and without compress, and to analyse the frequency of pressure ulcer occurrence and the intensity of this lesion.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1 month to 18 years old, according to the criteria of the paediatrics department of the Departmental Hospital la Roche sur Yon .
* Hospitalized in paediatrics ward or consultant in paediatric emergencies with a high probability of being hospitalized in paediatrics ward later.
* With an indication for the insertion of a short peripheral venous catheter
* Written agreement from the holder(s) of parental authority

Exclusion Criteria:

* Children with dermatological affections prior to inclusion and at the puncture site (atopic dermatitis, skin infection, skin wound, chickenpox, epidermolysis bullosa)
* Allergy to fixation devices
* Known immune deficient child
* Refusal of the patient or of the holders of parental authority to participate
* Life-saving emergency care
* Patient already included in the study
* Patient without social security coverage

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: stephanie Chaillot, Study Director — CHD VENDEE
Locations (1):
- CHD Vendee, La Roche-sur-Yon, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peripheral Venous Catheter With Compress | Peripheral Venous Catheter Without Compress
Started | 180 | 180
Completed | 136 | 137
Not Completed | 44 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peripheral Venous Catheter With Compress | Peripheral Venous Catheter Without Compress | Total
Number analyzed (Participants) | 180 | 180 | 360
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 11 [6.4 to 14.6] | 9.7 [4.5 to 13.8] | 10.5 [5.5 to 14.2]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One observation as a missing data about gender
  Participants
    number analyzed (Participants) | 180 | 179 | 359
    Female | 86 | 85 | 171
    Male | 94 | 94 | 188
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 180 | 180 | 360

OUTCOME MEASURES:

1. Primary Outcome: Pressure Ulcer of Grade >=1 on the National Pressure Ulcer Advisory Panel (NPUAP) Scale
Description: Occurrence of a pressure ulcer of grade ≥1 according to the NPUAP scale at the catheter extension junction. A higher grade on this scale indicates a worse patient outcome.
  The assessment will be performed in a blinded manner by a childcare assistant (CDA) from the department.
Time Frame: at catheter removal
Measure: Count of Participants; unit: Participants
Arm/Group | peripheral venous catheter with compress | peripheral venous catheter without compress
Number analyzed (Participants) | 136 | 137
Participants | 48 | 94

ADVERSE EVENTS:
Time Frame: Death, serious adverse events and other (non serious adverse events) were not assessed for the study
Description: Death, serious adverse events and other (non serious adverse events) were not assessed for the study
Arm/Group | Peripheral Venous Catheter With Compress | Peripheral Venous Catheter Without Compress
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT04540822/Prot_SAP_000.pdf